CLINICAL TRIAL: NCT04584632
Title: A Clinical Evaluation of the Efemoral Vascular Scaffold System (EVSS) for the Treatment of Patients with Symptomatic Peripheral Vascular Disease from Stenosis or Occlusion of the Femoropopliteal Artery
Brief Title: The Efemoral Vascular Scaffold System (EVSS) for the Treatment of Patients with Symptomatic Peripheral Vascular Disease from Stenosis or Occlusion of the Femoropopliteal Artery
Acronym: Efemoral I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efemoral Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL05122020
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease; Vascular Diseases; Stenosis; Femoropopliteal Stenosis
Keywords: Peripheral Artery Disease; Bioresorbable
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EVSS (Experimental): Efemoral Vascular Scaffold System (EVSS)
  Interventions: Device: Efemoral Vascular Scaffold System (EVSS)

INTERVENTIONS:
Device: Efemoral Vascular Scaffold System (EVSS) — Balloon-expandable, bioresorbable vascular scaffolds coated with sirolimus

SUMMARY:
To evaluate the safety and performance of the EVSS in patients with symptomatic peripheral vascular disease from stenosis or occlusion of the femoropopliteal artery

DETAILED DESCRIPTION:
The EFEMORAL I study is a prospective, single-arm, open-labeled, multi-center, clinical investigation enrolling patients with arterial diameter of ≥5.5 mm and ≤6.5 mm and lesion length ≤90 mm receiving a single EVSS.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral vascular occlusive disease (Rutherford-Becker Clinical Category 2-4)
* Patient with life expectancy >36 months
* Females of childbearing potential must have negative pregnancy test
* Patient is able to provide informed consent
* Patient agrees to undergo all protocol-required follow-up examinations and requirements at the investigational site.
* Patient must be able to take antiplatelet and/or anticoagulant agents as prescribed
* Single de novo native disease segment of the superficial femoral artery (SFA) or P1 popliteal segment
* Reference vessel diameter ≥5.5 mm and ≤6.5 mm
* Target lesion length ≤90 mm
* Target lesion with ≥50% DS
* Inflow artery and popliteal artery free from flow-limiting lesion (DS <50%)

Exclusion Criteria:

* Hemoglobin <9.0 g/dL
* WBC <3,000 cells/mm3
* Platelet count <80,000 cells/mm3 or >700,000 cells/mm3
* Acute or chronic renal dysfunction with creatinine >2.5 mg/dl (176 µmol/L)
* Severe liver impairment as defined by total bilirubin ≥3 mg/dl or two times increase over the normal level of SGOT or SGPT
* A known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, ticagrelor or sirolimus, or with contrast sensitivity for which the patient cannot be adequately pre-medicated
* Patient requires a planned procedure that would necessitate discontinuation of antiplatelet therapy
* Patient is unable to walk
* Patient has undergone a percutaneous vascular intervention <30 days prior to the planned index procedure
* Patient is maintained on chronic hemodialysis
* Patient has uncontrolled diabetes mellitus (HbA1c ≥7.0%).
* Patient has had a myocardial infarction within the previous 30 days of the planned index procedure
* Patient has had a stroke within the previous 30 days of the planned index procedure and/or has deficits from a prior stroke that limits the patient's ability to walk
* Patient has unstable angina defined as rest angina with ECG changes
* Patient has a local groin or acute systemic infection that has not been treated successfully or is currently under treatment
* Patient has acute thrombophlebitis, deep vein thrombosis or chronic venous insufficiency in either extremity
* Patient has other medical illnesses (e.g., cancer, congestive cardiomyopathy, etc.) that may cause the patient to be non-compliant with protocol requirements, confound the data interpretation or will prevent completion of all required follow up assessments through 36 months
* Patient is currently participating in an investigational drug, biologic, or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* Patient has ischemic or neuropathic ulcers on either foot
* Patient has undergone minor or major amputation of either lower extremity
* Patient is part of a vulnerable population who, in the judgment of the Investigator, is unable to give informed consent
* Target extremity with an angiographically significant (>50% DS) lesion located distal to the target lesion that requires treatment at the time of the index procedure or by a staged procedure
* Acute arterial ischemia of the target extremity
* Target extremity has been previously treated with open surgical revascularization (bypass or endarterectomy)
* Target vessel has been previously treated with stent, laser, atherectomy, surgical bypass, or endarterectomy
* Total occlusion (100% DS) of the ipsilateral inflow artery
* Angiographic evidence of thrombus in the target vessel
* The target lesion requires treatment with a device other than percutaneous transluminal balloon angioplasty (PTA) [e.g., orbital atherectomy, directional atherectomy, excimer laser, rotational atherectomy, cryoplasty, etc.]
* Target lesion is within or adjacent to an aneurysm
* Patient has angiographic evidence of thromboembolism or atheroembolism from treatment of an ipsilateral iliac lesion or from crossing or pre-dilating the target lesion
* Target lesion has moderate-to-severe calcification
* Target lesion with > 30% residual stenosis following pre-dilatation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Event (MAE) | 30 days
Freedom from Binary Restenosis | 12 months

SECONDARY OUTCOMES:
Device Success | Day 0
  Achievement of successful delivery and deployment of the study device(s) at the intended target lesion
Primary patency rate | 1, 6, 12, 24 and 36 months
Binary restenosis rate | 1, 6, 12, 24 and 36 months
Target lesion revascularization (TLR) | 1, 6, 12, 24 and 36 months
Ipsilateral extremity revascularization (IER) | 1, 6, 12, 24 and 36 months
Number of patients with Scaffold thrombosis | through 1 month
Number of patients with scaffold occlusion | 6, 12, 24 and 36 months
Rate of Major Adverse Limb Events | through 36 months
Ankle-brachial index (ABI) of target extremity | 1, 6, 12, 24 and 36 months
Limb salvage of target extremity | 1, 6, 12, 24 and 36 months
Rutherford-Becker Clinical Category for the target extremity | 1, 6, 12, 24 and 36 months
Walking impairment as assessed by Walking Impairment Questionnaire (WIQ) | 1, 6, 12, 24 and 36 months
Clinical Success | Up to 2 days after procedure
  Attainment of a final residual stenosis of <30% using the study device(s) and/or any adjunctive device at the intended target lesion without complications
Technical Success | Day 0
  Attainment of a final residual stenosis of <30% at the intended target lesion(

OTHER OUTCOMES:
Target lesion percent mean diameter stenosis | Post procedure (Day 0) and 6 months
Target lesion percent maximum diameter stenosis | post procedure (day 0) and at 6 months
Target lesion late lumen loss | 6 months
Ischemia-driven target lesion revascularization (IDTLR) | 1, 6, 12, 24 and 36 months
Amputation (minor and major) of the target extremity | 1, 6, 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Locations (4):
- Prince Of Wales Hospital, Sydney, Australia
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No